CLINICAL TRIAL: NCT01073865
Title: An Open Label, Randomised, Parallel Group, Multicentre Study to Compare ZOLADEX™ 10.8 mg Given Every 12 Weeks With ZOLADEX 3.6 mg Given Every 4 Weeks in Pre-menopausal Women With Oestrogen Receptor Positive Advanced Breast Cancer.
Brief Title: Study to Compare Zoladex™ 10.8 mg With Zoladex 3.6 mg in Pre-menopausal Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8666C00001
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
Keywords: ZOLADEX; Pre-menopausal; Oestrogen Receptor; Advanced Breast Cancer; Progression Free Survival
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Zoladex 10.8 mg (goserelin acetate) will be injected once every 12 weeks (± 7 days).
  One oral tamoxifen 20 mg tablet also will be taken daily
  Interventions: Drug: ZD9393 (Zoladex) 10.8 mg
- 2 (Active Comparator): Zoladex 3.6 mg (goserelin acetate) will be injected once every 4 weeks (± 7 days). One oral tamoxifen 20 mg tablet will also be taken daily.
  Interventions: Drug: ZD9393 (Zoladex) 3.6 mg

INTERVENTIONS:
Drug: ZD9393 (Zoladex) 10.8 mg — 10.8 mg (goserelin acetate): one subcutaneous depot injection once every 12 weeks (± 7 days).
  Other Names: Zoladex
  Arms: 1
Drug: ZD9393 (Zoladex) 3.6 mg — 3.6 mg (goserelin acetate): one subcutaneous depot injection once every 4 weeks (± 7 days).
  Other Names: Zoladex
  Arms: 2

SUMMARY:
The purpose of this study is to examine the efficacy and safety as well as the characteristics of the female hormone and study medications after administration in pre-menopausal women with estrogen receptor positive advanced breast cancer who were randomised in a 1:1 ratio to either of the two treatment groups; the ZD9393 3.6 mg depot group or ZD9393 10.8 mg depot group, both given in combination with tamoxifen tablets.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥20 years and pre-menopausal.Pre-menopausal defined as 1) last menses within 1 year of randomisation, and 2) E2 ≥10 pg/mL and FSH ≤ 30 mIU/mL within 4 weeks of randomisation.
* Hormone sensitivity (ER positive) of primary or secondary tumour tissue.
* Histological/cytological confirmation of breast cancer and are candidates to receive hormonal therapy as therapy for advanced breast cancer.

Exclusion Criteria:

* Patients who have received tamoxifen or other hormonal therapies as adjuvant therapy for breast cancer within 24 weeks before randomisation and/or who have received prior treatment with hormonal therapies for advanced breast cancer
* Patients who have received LHRHa as adjuvant therapy for breast cancer within 48 weeks before randomisation
* Patients who have relapsed during adjuvant hormonal therapy or within 48 weeks after completion of adjuvant hormonal therapy and/or

Ages: 20 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2010-02-26 (Actual); Primary Completion 2012-09-19 (Actual); Study Completion 2017-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Lindemann, PO, Study Director — AstraZeneca
Locations (42):
- India (11):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Chennai
  - Research Site, Hubli
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Mumbai
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Thiruvananthapuram
- Japan (17):
  - Research Site, Amagasaki-shi
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hamamatsu
  - Research Site, Hiroshima
  - Research Site, Kagoshima
  - Research Site, Kamogawa-shi
  - Research Site, Kitaadachi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mitaka-shi
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Sapporo
- Philippines (5):
  - Research Site, Cebu City
  - Research Site, Iloilo City
  - Research Site, Lipa City
  - Research Site, Pasay
  - Research Site, Quezon City
- South Korea (2):
  - Research Site, Seoul
  - Research Site, Suwon
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Maharat Nakorn Ratchasima
  - Research Site, Songkhla
  - Research Site, Ubonratchathani

REFERENCES:
- See also: D8666C00001ClinicalStudyProtocol_personal_info_redacted_12December.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=637&filename=D8666C00001ClinicalStudyProtocol_personal_info_redacted_12December.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Totally 286 patients were screened to the study from 58 centres in the following 6 countries: India, Japan, Korea, Philippines, Thailand, Taiwan. The first patient entered the study on 26 February 2010 and the last visit of last patient was on 19 September 2012.
Pre-assignment Details: 286 patients were screened and 222 patients were randomized (109 in ZOLADEX 10.8 mg, 113 in ZOLADEX 3.6 mg)
Groups:
- Zoladex 10.8 mg: ZOLADEX 10.8 mg (goserelin acetate): one subcutaneous depot injection into interior abdominal wall once every 12 weeks
- Zoladex 3.6 mg: ZOLADEX 3.6 mg (goserelin acetate): one subcutaneous depot injection into interior abdominal wall once every 4 weeks
Period: Overall Study
Arm/Group | Zoladex 10.8 mg | Zoladex 3.6 mg
Started | 109 (Number of patients randomised) | 113 (Number of patients randomised)
Received Randomised Treatment | 108 (Number of patients received randomised treatment) | 113 (Number of patients received randomised treatment)
Completed | 81 (Number of patients completed the study) | 74 (Number of patients completed the study)
Not Completed | 28 | 39
Not completed — Reasons other than below | 19 | 31
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoladex 10.8 mg | Zoladex 3.6 mg | Total
Number analyzed (Participants) | 109 | 113 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (6.9) | 40.9 (6.0) | 40.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 113 | 222
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 109 | 113 | 222
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 109 | 113 | 222
  Other | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Asia: India | 29 | 27 | 56
  Asia: Japan | 29 | 30 | 59
  Asia: Philippines | 21 | 23 | 44
  Asia: Thailand | 10 | 9 | 19
  Asia: Taiwan | 7 | 9 | 16
  Asia: Republic of Korea | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Progression-free Survival (PFS) at 24 Weeks
Description: A patient is judged as progression-free survive at Week 24 if their PFS time is at least 24 weeks with no progression event prior to Week 24 (ie, overall visit response is complete response (CR), partial response (PR) or stable disease (SD) at a tumour assessment at least 24 weeks after randomization). Overall visit response is assessed according to the RECIST version 1.1. %PFS is the proportion of patients with PFS.
Time Frame: 24 weeks after the first dosing
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Zoladex 10.8 mg | Zoladex 3.6 mg
Number analyzed (Participants) | 109 | 113
Participants | 67 | 68
Statistical Analysis 1: Comparison: Zoladex 10.8 mg vs Zoladex 3.6 mg; CI for the difference (10.8 mg-3.6 mg) in %PFS at 24 weeks calculated using the score method recommended by Newcombe et al; Test type: Non-Inferiority or Equivalence — The lower limit of the CI of the difference is greater than or equal to -17.5%. This non-inferiority margin was pre-defined in the study protocol; Risk Difference (RD) = 1.29, 95% CI 2-sided [-11.40 to 13.90] — %PFS at 24 weeks for Zoladex 10.8mg - %PFS at 24 weeks for Zoladex 3.6mg

2. Secondary Outcome: Number of Responders at 24 Weeks
Description: Responders are defined as those patients with a best objective tumour response of CR or PR during the first 24 weeks of therapy. Tumour response is assessed according to the RECIST version 1.1. ORR is defined as the proportion of patients who are responders.
Time Frame: 24 weeks after the first dosing
Population: Full Analysis Set (patients without measurable disease at baseline were excluded from analysis)
Measure: Count of Participants; unit: Participants
Arm/Group | Zoladex 10.8 mg | Zoladex 3.6 mg
Number analyzed (Participants) | 88 | 93
Participants | 21 | 25
Statistical Analysis 1: Comparison: Zoladex 10.8 mg vs Zoladex 3.6 mg; CI for the difference (10.8 mg-3.6 mg) in ORR at 24 weeks calculated using the score method recommended by Newcombe et al; Test type: Superiority or Other; Risk Difference (RD) = -3.02, 95% CI 2-sided [-15.47 to 9.67] — ORR at 24 weeks for Zoladex 10.8mg - ORR at 24 weeks for Zoladex 3.6mg

3. Secondary Outcome: Oestradiol (E2) Serum Concentrations at 24 Weeks
Description: E2 serum concentrations (pg/mL) at 24 weeks
Time Frame: 24 weeks after the first dosing
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Zoladex 10.8 mg | Zoladex 3.6 mg
Number analyzed (Participants) | 74 | 70
pg/mL | 20.302 (12.251) | 24.798 (28.149)

ADVERSE EVENTS:
Time Frame: Non serious AEs and SAEs were be collected from the time of patient informed until 4 weeks after the final administration of ZOLADEX 3.6 mg or 12 weeks after the final administration of ZOLADEX 10.8 mg
Arm/Group | Zoladex 10.8 mg | Zoladex 3.6 mg
All-Cause Mortality (participants affected / at risk) | 4/108 | 3/113
Serious Adverse Events (participants affected / at risk) | 4/108 | 8/113
Other Adverse Events (participants affected / at risk) | 47/108 | 52/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoladex 10.8 mg (N=108) | Zoladex 3.6 mg (N=113)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PERIODONTAL DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
TETANUS (Infections and infestations) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoladex 10.8 mg (N=108) | Zoladex 3.6 mg (N=113)
HOT FLUSH (Vascular disorders) | 15 | 22
NASOPHARYNGITIS (Infections and infestations) | 13 | 9
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 9
HEADACHE (Nervous system disorders) | 7 | 7
NAUSEA (Gastrointestinal disorders) | 2 | 9
CONSTIPATION (Gastrointestinal disorders) | 4 | 5
VOMITING (Gastrointestinal disorders) | 4 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 4
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 5
PYREXIA (General disorders) | 2 | 7
FATIGUE (General disorders) | 1 | 4
INSOMNIA (Psychiatric disorders) | 3 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 4
ANAEMIA (Blood and lymphatic system disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs cannot disclose trial results without prior approval in writing by the sponsor.